CLINICAL TRIAL: NCT02873949
Title: Analysis of Soluble TREM (Triggering Receptor Expressed on Myeloid Cells)-1 and -2 in Crevicular Fluid and Associated Bacterial Flora in Patients Affected by Periodontitis
Acronym: TREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A00097-44
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Periodontitis
Keywords: immunology factors; TREM; stress
MeSH Terms: conditions — Periodontitis | interventions — Psychometrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Periodontitis patients (Other): 30 patients consulting at Odontology department for periodontal treatment
  Interventions: Biological: Crevicular samples (1-10µl); Biological: Saliva samples (1ml); Other: Etiologic treatment; Other: Psychometric tests
- 2. Control (Other): 10 patients not affected by periodontitis consulting at Odontology department for checkup of teeth state and/or scaling
  Interventions: Biological: Crevicular samples (1-10µl); Biological: Saliva samples (1ml); Other: Psychometric tests

INTERVENTIONS:
Biological: Crevicular samples (1-10µl) — In periodontitis patients: from 2 sites affected by periodontitis and 1 healthy site, 2 samples/site, before and after treatment
  In non-periodontitis individuals: 2 samples from 1 site
Biological: Saliva samples (1ml)
Other: Etiologic treatment — education on oral hygiene, scaling and root planing
  Arms: 1. Periodontitis patients
Other: Psychometric tests — Spielberger State-Trait Anxiety Inventory and Cohen Perceived Stress Scale

SUMMARY:
Etiopathology of periodontitis is complex and various risk factors are known :

* Bacterial factors: major risk factor. Although the presence of periodontopathogen bacteria is necessary for the onset of periodontitis, these microorganisms are not sufficient for progression of all periodontal disease.
* Immune factor: host immune response modulates the disease evolution to destruction or recovery. The most studied cytokine in periodontology is IL-1 that induces various immune reactions and bone resorption directly or indirectly through the stimulation of prostaglandin E2 (PGE2) release. PGE2 activates the matrix metalloproteinases that are responsible of the degradation of bone extracellular matrix.

Cytokine production, especially TNFα, IL-1β, IL-6 and IL-8, by some immune cells is modulated by new identified molecules such as Triggering Receptor Expressed on Myeloid cells (TREM) whose role in periodontitis is unknown.

The purpose of this study is to compare concentrations of soluble TREM-1 and TREM-2 markers in infected sites and in healthy sites in patients affected by periodontitis.

Other purposes are

1. Comparison of soluble TREM-1 and TREM-2 concentrations in healthy sites in patients affected by periodontitis and in healthy patients
2. Comparison of soluble TREM-1 and TREM-2 concentrations before and after etiologic periodontitis treatment
3. Estimation of the correlation between soluble TREM-1 and TREM-2 concentrations and clinical signs of periodontitis
4. Description of soluble TREM-1/TREM-2 ratio before and after etiologic treatment
5. Description of presence of some bacteria in sites analyzed for soluble TREM-1 and TREM-2
6. Search for the most observed bacteria in presence of high concentrations of soluble TREM-1 and TREM-2 before and after etiologic treatment
7. Evaluation of the impact of psychological stress measured through salivary cortisol level in saliva on TREM-1 and -2 expression
8. Evaluation of the impact of psychological stress through stress and anxiety auto-questionnaires (Spielberger and Cohen) on soluble TREM-1 and TREM-2 concentrations in crevicular fluid of healthy and pathologic teeth.

ELIGIBILITY:
Inclusion Criteria:

All:

* Affiliation to social security plan
* Absence of refusal of patient

Group 1. Periodontal patients:

* Affected by moderate to severe chronic periodontitis
* At least 2 distinct infected sites with periodontal pocket depth ≥ 5mm
* Having not received any root planing during last 6 months before visit

Group 2. Control:

* No periodontitis
* Consulting for dental checkup and eventually scaling

Exclusion Criteria:

All:

* Pregnant women (change in bacterial flora) and breast-feeding
* Administration of systemic antibiotherapy or any treatment influencing periodontal environment (anti-inflammatory, anti-epileptic, immune-suppressor, calcium inhibitor) during 6 months before sample collection
* Patients having a pathology needing a prophylactic antibiotherapy (possibly influencing the treatment)
* Teeth with periapical inflammatory lesions of endodontic origin
* Person under guardianship

Group 1. Periodontal patients:

- Root planing during last 6 months before visit

Group 2. Control:

- Periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Average concentration (quantified with ELISA assay) of soluble TREM-1 and TREM-2 in crevicular fluid from 2 distant sites affected by periodontitis and 1 healthy site of each periodontitis patients at first consultation | day 0

SECONDARY OUTCOMES:
Average concentration (quantified with ELISA assay) of soluble TREM-1 and TREM-2 in crevicular fluid from healthy sites of periodontitis patients and non-periodontitis patients at first consultation | day 0
  Crevicular fluid from 3 sites (2 distant affected by periodontitis and 1 healthy) of periodontitis patients and from 1 healthy site of non-periodontitis patients
Average concentration (quantified with ELISA assay) of soluble TREM-1 and TREM-2 in crevicular fluid of periodontitis patients before and after etiologic treatment of periodontitis | day 0 and after 13 to 15 weeks (after etiologic treatment of periodontitis patients)
  Crevicular fluid from 3 sites (2 distant affected by periodontitis and 1 healthy) of periodontitis patients
Identification of periodontal bacterial flora | day 0 and after 13 to 15 weeks (after etiologic treatment of periodontitis patients)
  The kit microIDent®plus11 (Hain, Lifesciences) allows the identification by PCR of the most pathogen periodontal bacteria.
Psychological stress score with Cohen Perceived Stress Scale | day 0
Psychological stress score with Spielberger State-Trait Anxiety Inventory | day 0
Quantification of salivary cortisol by ELISA to measure psychological stress | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BISSON, Principal Investigator — Service Odontologie - Site Heydenreich - CHRU Nancy; Sébastien GIBOT, Study Chair — Service Réanimation Médicale - Hôpital Central - CHRU Nancy
Locations (1):
- Service Odontologie - Site Heydenreich - CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No